CLINICAL TRIAL: NCT00680355
Title: Bioavailability of Golden Rice Carotenoids in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Guangwen Tang, Ph. D, Senior Scientist, Tufts University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 59-1956-6-656
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: golden rice carotenoids; healthy volunteers; retinol equivalence
MeSH Terms: interventions — Corn Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Golden rice meal with 10g fat (Other): 10 g corn oil in the Golden Rice meal
  Interventions: Dietary Supplement: golden rice; Dietary Supplement: corn oil 10g
- Golden Rice with 0g fat (Other): 0g corn oil eating with the Golden Rice meal
  Interventions: Dietary Supplement: golden rice; Dietary Supplement: corn oil 0g
- Golden Rice meal with 5 g fat (Other): 5 g corn oil in the Golden Rice meal
  Interventions: Dietary Supplement: golden rice; Dietary Supplement: coren oil 5 g

INTERVENTIONS:
Dietary Supplement: golden rice — An acute dose of cooked golden rice containing ~ 1 mg of ß-carotene
  Other Names: golden rice carotenoids
Dietary Supplement: corn oil 0g — 0 g of corn oil in the golden rice meal
  Arms: Golden Rice with 0g fat
Dietary Supplement: corn oil 10g — 10g corn oil in the golden rice meal
  Arms: Golden rice meal with 10g fat
Dietary Supplement: coren oil 5 g — golden rice meal with 5 g corn oil
  Arms: Golden Rice meal with 5 g fat

SUMMARY:
This investigation protocol uses an isotope reference method to evaluate bioavailability of ß-C in rice and its bioconversion to vitamin A.

A well-nourished population will be fed hydroponically grown Golden Rice containing ~ 1 mg of β-carotene at day 8 after a reference dose of vitamin A at day 1. The blood samples will be collected up to 33 days after the doses. The absorption kinetics will be determined by tracking both vitamin A and β-carotene in human serum. Blood responses to Golden Rice β-carotene will be determined and evaluated. The vitamin A value of Golden Rice can thus be quantitatively determined.

DETAILED DESCRIPTION:
Recently, scientists have genetically engineered "golden rice" that contains 1.6 ug ß-carotene in a gram of dry rice (12). Since the vitamin A equivalency varies from 2 ug (oil dose) to 27 ug (vegetable) carotene to 1 retinol equivalent and the equivalency is matrix dependent, it is necessary to know what the vitamin A equivalency of golden rice beta-carotene is. The determination of the absorption and conversion of golden rice beta-carotene is of importance for designing food programs in many rice-eating regions of the world, where vitamin A deficiency is common.

To evaluate the absorption and intestinal conversion of rice beta-carotene after an acute dose of golden rice, an intrinsically labeled Golden Rice with a labeled reference dose of vitamin A are used. We propose to conduct a pilot study on the US adults with normal vitamin A status (n = 15).

The specific aims of this pilot study are:

1. To determine ß-carotene response kinetics following a meal of golden rice with 0, 5, or 10 g fat (butter);
2. To determine retinol kinetics from the golden rice and from the labeled vitamin A dose;
3. To determine vitamin A value of golden rice ß-carotene in adults with normal vitamin A status. The determination of the absorption and conversion of golden rice ß-carotene is of importance for designing food programs in many rice-eating regions of the world, where vitamin A deficiency is common.

ELIGIBILITY:
Inclusion Criteria:

* healthy health

Exclusion Criteria:

* GI track problems

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The enrichment of labeled golden rice β-carotene and its conversion to labeled retinol in serum samples after the golden rice meal with 0, 5, or 10 g fat (butter) as compared to the reference dose of vitamin A that is labeled differently. | 33 days

CONTACTS AND LOCATIONS:
Overall Officials: Guangwen Tang, Ph. D, Principal Investigator — Tufts University
Locations (1):
- USDA Human Nutrition Research Center on Aging at Tufts Uni, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Tang G, Qin J, Dolnikowski GG, Russell RM, Grusak MA. Golden Rice is an effective source of vitamin A. Am J Clin Nutr. 2009 Jun;89(6):1776-83. doi: 10.3945/ajcn.2008.27119. Epub 2009 Apr 15. PMID 19369372